CLINICAL TRIAL: NCT03407300
Title: A Prospective, Randomized Clinical Study of Safety and Efficacy by Using Docetaxel With or Without Traditional Chinese Medicine XH1 in Patients With Stage ⅢB-Ⅳ Non-small Cell Lung Cancer (NSCLC) Who Failed With First-line Chemotherapy
Brief Title: A Safety and Efficacy Trial of Docetaxel With or Without XH1 in Non-small Cell Lung Cancer (NSCLC) Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haining Health-Coming Biotech Co., Ltd. (Other)
Collaborators: Alphacait, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Alphacait-XH1-201711
Record Dates: First submitted 2018-01-12; First posted 2018-01-23 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Non-small Cell Lung Cancer (NSCLC), XH1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Docetaxel (Active Comparator): Stage III-IV NSCLC patients who failed first-line chemotherapy will be treated with Docetaxel alone.
  Interventions: Drug: Docetaxel
- Docetaxel plus XH1 (Active Comparator): Stage III-IV NSCLC patients who failed first-line chemotherapy will be treated with Docetaxel plus Chinese traditional medicine XH1.
  Interventions: Drug: Docetaxel; Drug: Chinese traditional medicine XH1

INTERVENTIONS:
Drug: Docetaxel — To evaluate the safety and efficacy of Docetaxel alone in stage III-IV NSCLC patients
Drug: Chinese traditional medicine XH1 — To evaluate the safety and efficacy of Docetaxel combined with Chinese tradition medicine XH1 in stage III-IV NSCLC patients
  Arms: Docetaxel plus XH1

SUMMARY:
This is a prospective, randomized, multicenter clinical study designed to evaluate its safety and efficacy by using Docetaxel with or without Traditional Chinese Medicine XH1 in patients with Stage ⅢB-Ⅳ Non-small Cell Lung Cancer (NSCLC) who failed with first-line Chemotherapy. The primary outcome measure includes progression-free survival (PFS) after treatment. Secondary outcome measures include collecting biomarkers before and during treatment, overall survival (OS), objective response rate (ORR), disease control rate (DCR), and patient's quality of life.

DETAILED DESCRIPTION:
Lung cancer is one of the most common malignant tumors in the world and has become the No. 1 cause of death from malignant tumors in China. Non-small cell lung cancer (NSCLC) includes squamous cell carcinomas, adenocarcinomas, and large cell carcinomas and accounts for about 80-85% of all lung cancers. NSCLC cancer cells divide slowly in a diffusive manner and metastasize at a relatively late stage compared to small cell carcinomas. A majority of patients with NSCLC are already in advanced stages and have a low 5-year survival rate.

Treatments for advanced NSCLC include chemotherapy and targeted therapies. Platinum is currently used in the first-line treatment combination with Pemetrexed / gemcitabine / docetaxel / paclitaxel / vinorelbine and etc. For EGFR mutation negative patients, chemotherapy remains to be the preferred treatment of choice. Selection of chemotherapy regimes should take full account of patient's condition, including patient's physical condition. Assessments regarding patient's possible benefits from chemotherapy should include timely evaluation of efficacies, close observation of adverse events and effective control of adverse reactions. Traditional Chinese Medicine (TCM) has in recent years become an important adjunct for lung cancer treatment. TCM has been shown to be effective in stabilizing the tumor, prolonging patient survival, increasing immune function, improving clinical symptoms, improving quality of life and reducing the adverse events of radiotherapy and chemotherapy.

With the advent of new technologies, TCM has been shown to have a variety of therapeutic effects towards multiple tumor-associated genes. However, it remains a major obstacle as to how to effectively screen and select TCM remedies that are effective against lung cancer and meet the efficacy standards of contemporary cancer care.

Under the premises described above, investigators developed a novel drug screening and selection model (Alphacait) in tumor microenvironment using Synthetic Lethal and accelerated RNA Speedup PDX aided by artificial intelligence calculation. This model could provide new treatment options for patients with EGFR negative late-stage lung cancer through conducting synthetic lethal analysis in vitro and in vivo using patient's own cancer cells and selecting the most effective combination therapies for these patients. As this approach aims at selecting individualized medications for a specific patient using patient's own cancer cells, it enables rapid exclusion of false positives and accurate determination of potentially effective treatment regimens for each individual patient.

The Alphacait model thus involves acquisition of patient's cancer cells through biopsy, combinatorial chemistry techniques, cancer cell culture in vitro, and cancer cell transplantation and growth in vivo in a microenvironment similar to that in a living human body. Using this model, investigators will be able to screen thousands of different TCM combinations in a matter of days. The inhibitory curves of the Synthetic Lethal RNA expression for each drug combination specific to a patient's cancer cells could be obtained within 72 hours to determine the most promising anticancer drug combinations. The cancer cells will thereafter be transplanted into immune deficient rats for further testing and validation in vivo in a living microenvironment. Investigators expect to complete the screening experiments in vitro and validation experiments in vivo within 6 weeks of biopsy and select the most effective drug combinations. This information is then conveyed to the clinicians to guide the selection of therapeutic regimes involving TCM in conjunction with patient's preferences and clinician's experiences.

Investigators have screened a total of 250,000 drug combinations using the Alphacait model and determined that approximately 100 drugs may be useful against NSCLC cancer cells. Preliminary testing of the model in about 200 patients in China found that the TCM combination XH1 plus docetaxel were effective in a subgroup of patients with end-stage NSCLC. The aim of the present study is to further confirm the efficacy of this combination in a randomized and controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically diagnosed IIIB or IV non-small cell lung cancer and EGFR negative
2. Previously accepted first-line standard treatment failure or recurrence
3. At least one measurable lesion
4. From the last radiotherapy interval of at least 4 weeks, recovery from acute toxicity of radiation, prophylactic brain radiotherapy or palliative bone metastases lesions except radiotherapy
5. Any gender, age ≥18 years
6. ECOG PS : 0-2 points
7. Expected survival ≥ March
8. The level of organ function meets the following criteria (1) subject to the standard blood test: ANC ≥ 1.5 × 10 9 / L, PLT ≥ 8 0 × 10 9 / L, Hb ≥ 100 g / L (2) biochemical tests must meet the following criteria: TBIL <1.5 × U LN, ALT, AST <2 .5 × ULN ( if liver ALT, AST can be <5 × U LN), BUN, and Cr ≤ 1 × ULN)
9. Patients must be willing to eight weeks after the use of appropriate methods of contraception and the last administration of the test drug during the test, or surgically sterile
10. Subjects volunteered to join the study, signed informed consent, good compliance, with follow-up

Exclusion Criteria:

1. Symptomatic brain metastasis (could still enroll into the study if treatment finished 21 days prior to the enrollment and the patient is stable, but brain MRI, CT or angiogram is needed to rule out no intracranial hemorrhage)
2. Following cardiac disease: second-degree or above cardiac ischemia or myocardial infarction, uncontrolled arrhythmias (including QTc interval male>450 ms, female>470ms), according to NYHA criteria, III to IV cardiac insufficiency, or echocardiogram reveals left ventricular ejection fraction (LVEF) <50%
3. History of pulmonary interstitial lung disease or active interstitial lung disease;
4. Coagulation dysfunction (INR >1.5 or PT>ULN+ 4sec, or PTT>1.5 ULN), with bleeding tendency or currently receiving thrombolysis therapy or anticoagulation treatment;
5. Major surgery, severe traumata, fracture or ulcers within past 4 weeks.
6. Active infections requiring antimicrobial therapy (e.g., requires the use of antimicrobial drugs, antiviral, antifungal therapy)
7. Participation of other cancer chemotherapy clinical study within past 4 weeks;
8. History of uncured coexisting cancer, not including cured basal cell carcinoma, cervical cancer in situ, or superficial bladder cancer
9. Pregnant or breast feeding women; fertile patients not willing or able to take effective contraceptive measures
10. Any circumstances that might affect the proceeding of the clinical trial and/or research result analysis, as determined by the clinical investigator(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 12 month
  Time from randomization until disease progression or death

SECONDARY OUTCOMES:
Overall survival (OS) | 12month
  Time from randomization until death from any cause
Objective response rate (ORR) | 12 month
  Proportion of patients with reduction in tumor burden of a predefined amount
Disease control rate (DCR) | 12 month
  The sum of complete responses (CR) + partial responses (PR) + stable disease (SD)
Incidence of Treatment-Emergent Adverse Events | 12 month
  Drug-related adverse reactions including SAE and AE must be recorded, mainly in the following： Severe cardiovascular, pulmonary, liver and kidney damage; myelosuppression including neutropenia, anemia and thrombocytopenia; muscle fatigue, pain, imbalance; Oral ulcers: the patient's gums, cheeks, throat and tongue are prone to ulcers; nausea, vomiting, constipation or diarrhea; hair loss; skin discomfort; hormonal fluctuations, anxiety and depression.

OTHER OUTCOMES:
Biomarkers | 12 months
  Using Next Generation Sequencing (NGS), Nanostring technology to assess the presence of newly diagnosed and / or newly acquired tumor tissue and its response to disease states and / or therapies Relevance, and explore the correlation between the status of the biomarkers and the response to treatment before and during treatment.
  The list of biomarkers: CEA, SCC, NSE, Cyfra 21-1, CA125, ProGRP

CONTACTS AND LOCATIONS:
Overall Officials: Enguo Chen, MD, Principal Investigator — Sir Run Run Shaw Hospital; Haizhou Lou, MD, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Through publication after study completion
Supporting Information: Study Protocol, CSR
Time Frame: June, 2019